CLINICAL TRIAL: NCT00892775
Title: Immunogenicity & Safety Study of GSK Biologicals' 208136 Vaccine Formulated With New Measles and Rubella Working Seeds
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 108760; 2011-005881-38 (EudraCT Number)
Record Dates: First submitted 2009-05-04; First posted 2009-05-05 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Measles; Varicella; Mumps; Rubella
Keywords: Working seed virus; Rubella; Mumps; Varicella; Combined measles-mumps-rubella-varicella vaccine; Pediatric immunization; Measles
MeSH Terms: conditions — Measles; Chickenpox; Mumps; Rubella

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Priorix-Tetra new WS Group (Experimental): Subjects received 2 doses of Priorix-Tetra vaccine formulated with new measles and rubella working seeds at Day 0 and Week 12.
  Interventions: Biological: GSK Biologicals' 208136, new formulation
- Priorix-Tetra current WS Group (Experimental): Subjects received 2 doses of Priorix-Tetra vaccine manufactured with current working seed virus at Day 0 and Week 12.
  Interventions: Biological: Priorix-Tetra (combined measles-mumps-rubella-varicella vaccine)

INTERVENTIONS:
Biological: Priorix-Tetra (combined measles-mumps-rubella-varicella vaccine) — Vaccine will be administered subcutaneously in the left upper arm (deltoid region)
  Arms: Priorix-Tetra current WS Group
Biological: GSK Biologicals' 208136, new formulation — Vaccine will be administered subcutaneously in the left upper arm (deltoid region)
  Arms: Priorix-Tetra new WS Group

SUMMARY:
This study is undertaken to generate clinical data on GSK Biologicals' combined measles-mumps-rubella-varicella vaccine manufactured with measles and rubella obtained from newly established working seed viruses which are one passage further than the current working seed viruses. The measles-mumps-rubella-varicella vaccine manufactured with the current working seed viruses will serve as comparator.

A seed lot system is a system according to which successive batches of a vaccine are derived from the same master seed virus. For routine production, a working seed lot is prepared from the master seed virus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* A male or female between, and including, 11 and 21 months of age (e.g. from age 11months until the day before age 22 months) at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject after they have been advised on the risks and benefits of the study in a language they clearly understand, and before performance of any study procedure.
* Free of obvious healthy problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Administration of immunoglobulins and/or any blood products during the six months before entering the study or planned administration during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within 30 days prior to until 42 days after each study vaccine dose with the exception of oral polio vaccine (OPV) which can be given at any time and routine inactivated vaccines such as pneumococcal, meningococcal or Haemophilus influenzae type b conjugate vaccines, inactivated influenza or diphtheria/tetanus containing vaccines which can be administered up to eight days before each study vaccine dose.
* Previous vaccination against measles, mumps, rubella and/or varicella.
* History of measles, mumps, rubella and/or varicella/zoster diseases.
* Known exposure to measles, mumps, rubella and/or varicella within 30 days prior to study start.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s), including systemic hypersensitivity to neomycin.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Rectal temperature ≥38°C or axillary temperature >=37.5°C at the time of vaccination.
* Residence in the same household as a high risk person e.g.:
* New-born infants (0-4 weeks of age)
* Pregnant women who have a negative history of chickenpox
* Persons with known immunodeficiency

Ages: 11 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 501 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2010-09-17 (Actual); Study Completion 2010-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Singapore, Singapore
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Huang LM, Lee BW, Chan PC, Povey M, Henry O. Immunogenicity and safety of combined measles-mumps-rubella-varicella vaccine using new measles and rubella working seeds in healthy children in Taiwan and Singapore: a phase II, randomized, double-blind trial. Hum Vaccin Immunother. 2013 Jun;9(6):1308-15. doi: 10.4161/hv.24035. Epub 2013 Feb 20. PMID 23425607
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 108760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108760 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 501 enrolled participants, 3 were not administered any vaccine and hence were not considered as having started the study.
Period: Overall Study
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Started | 332 | 166
Completed | 327 | 165
Not Completed | 5 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Subject difficulties with blood drawing | 1 | 0
Not completed — Disclaimer/ Withdrawal caused by H1N1 | 1 | 0
Not completed — Migrated/ moved from study area | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group | Total
Number analyzed (Participants) | 332 | 166 | 498
Age, Continuous [Mean (Standard Deviation); unit: Months] | 13 (1.94) | 12.9 (1.7) | 12.97 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 84 | 250
  Male | 166 | 82 | 248
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian heritage | 165 | 83 | 248
  Asian - South East Asian heritage | 162 | 81 | 243
  White - Caucasian / European heritage | 3 | 1 | 4
  Unspecified | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Seroconverted for Measles, Mumps, Rubella and Varicella Antibodies Greater Than or Equal to (≥) the Cut-off Value.
Description: Seroconversion was defined as the appearance of antibodies in the serum of subjects seronegative before vaccination. The cut-off values for seroconversion was 150 milli international units per milliliter (mIU/mL), 231 units per milliliter (U/mL), 4 international units per milliliter (IU/mL) and 1:4 dilution for measles, mumps, rubella and varicella, respectively.
Time Frame: At 42-56 days after the first dose of study vaccine (Week 6)
Population: The According-to-protocol (ATP) cohort for immunogenicity included all eligible subjects who were seronegative at baseline to at least one vaccine antigen, who had received vaccine according to their random assignment, who had not received a vaccine forbidden in the protocol and for whom pre/ post-vaccination serology results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 314 | 157
Participants
  Anti-measles ≥ 150 mIU/mL | 312 | 157
  Anti-mumps ≥ 231 U/ML | 279 | 142
  Anti-rubella ≥ 4 IU/mL | 313 | 157
  IgG varicella antibodies ≥ 1:4 dilution | 284 | 131
Statistical Analysis 1: Comparison: Priorix-Tetra New WS Group vs Priorix-Tetra Current WS Group; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for measles 42-56 days after vaccination was concluded if the lower limit of the 95% confidence interval around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = -0.64, 95% CI 2-sided [-2.29 to 1.76]
Statistical Analysis 2: Comparison: Priorix-Tetra New WS Group vs Priorix-Tetra Current WS Group; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for mumps 42-56 days after vaccination was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = -0.74, 95% CI 2-sided [-6.14 to 5.58]
Statistical Analysis 3: Comparison: Priorix-Tetra New WS Group vs Priorix-Tetra Current WS Group; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for rubella 42-56 days after vaccination was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = -0.32, 95% CI 2-sided [-1.78 to 2.08]
Statistical Analysis 4: Comparison: Priorix-Tetra New WS Group vs Priorix-Tetra Current WS Group; Test type: Non-Inferiority — Non-inferiority with respect to seroconversion rates for varicella 42-56 days after vaccination was concluded if the lower limit of the 95% CI around the difference in seroconversion rates between groups would be [-10%] or higher; Difference in percentage = 4.69, 95% CI 2-sided [0.72 to 10.34]

2. Secondary Outcome: Number of Subjects Seroconverted for Measles, Mumps, Rubella and Varicella Antibodies ≥ the Cut-off Value.
Description: Seroconversion was defined as the appearance of antibodies in the serum of subjects seronegative before vaccination. The cut-off values for seroconversion was 150 mIU/mL, 231 U/mL, 4 IU/mL and 1:4 dilution for measles, mumps, rubella and varicella, respectively.
Time Frame: At 42-56 days after the second dose of study vaccine (Week 18)
Population: The ATP cohort for immunogenicity included all eligible subjects who were seronegative at baseline to at least one vaccine antigen, who had received the comparator vaccine according to their random assignment, who had not received a vaccine not specified/ forbidden in the protocol and for whom pre/ post-vaccination serology results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 308 | 156
Participants
  Anti-measles ≥ 150 mIU/mL | 308 | 156
  Anti-mumps ≥ 231 U/ML | 307 | 155
  Anti-rubella ≥ 4 IU/mL | 308 | 156
  IgG varicella antibodies ≥ 1:4 dilution | 286 | 138

3. Secondary Outcome: Antibody Titers Against Measles, Mumps, Rubella and Varicella Viruses
Description: Antibody titers were summarized by geometric mean titers (GMTs) with their 95% confidence intervals.
Time Frame: At 42-56 days after the first and second dose of study vaccine(s).
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 314 | 157
Titres
  Anti-Measles (mIU/mL); Dose 1 | 3291.2 [3054 to 3546.8] | 3460.1 [3145.6 to 3806]
  Anti-Mumps (U/mL); Dose 1: number analyzed (Participants) | 311 | 157
  Anti-Mumps (U/mL); Dose 1 | 924.4 [821.9 to 1039.7] | 994.4 [851.7 to 1161]
  Anti-Rubella (IU/mL); Dose 1 | 71.7 [66.1 to 77.9] | 66.6 [59.3 to 74.9]
  Anti-Varicella (1/dil); Dose 1: number analyzed (Participants) | 291 | 141
  Anti-Varicella (1/dil); Dose 1 | 104.8 [90.8 to 120.9] | 69.6 [53.6 to 90.2]
  Anti-Measles (mIU/mL); Dose 2: number analyzed (Participants) | 308 | 156
  Anti-Measles (mIU/mL); Dose 2 | 4247.6 [3911.5 to 4612.6] | 4297.1 [3867.9 to 4774]
  Anti-Mumps (U/mL); Dose 2: number analyzed (Participants) | 307 | 155
  Anti-Mumps (U/mL); Dose 2 | 3379.5 [3121.3 to 3659] | 3216.2 [2870.9 to 3603]
  Anti-Rubella (IU/mL); Dose 2: number analyzed (Participants) | 308 | 156
  Anti-Rubella (IU/mL); Dose 2 | 125.7 [117.4 to 134.5] | 115.2 [104.2 to 127.4]
  Anti-Varicella (1/dil); Dose 2: number analyzed (Participants) | 286 | 138
  Anti-Varicella (1/dil); Dose 2 | 6570.6 [5746.7 to 7512.7] | 5134.8 [4153.8 to 6347.4]

4. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/ spontaneously painful. Grade 3 redness/ swelling = redness/ swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: Within 4 days after each vaccination (Days 0-3)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects, with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 330 | 166
Participants
  Any Pain; Dose 1 | 62 | 28
  Grade 3 Pain; Dose 1 | 0 | 0
  Any Redness; Dose 1 | 92 | 44
  Grade 3 Redness; Dose 1 | 2 | 3
  Any Swelling; Dose 1 | 22 | 11
  Grade 3 Swelling; Dose 1 | 0 | 0
  Any Pain; Dose 2: number analyzed (Participants) | 327 | 164
  Any Pain; Dose 2 | 46 | 24
  Grade 3 Pain; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 Pain; Dose 2 | 0 | 0
  Any Redness; Dose 2: number analyzed (Participants) | 327 | 164
  Any Redness; Dose 2 | 79 | 43
  Grade 3 Redness; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 Redness; Dose 2 | 4 | 5
  Any Swelling; Dose 2: number analyzed (Participants) | 327 | 164
  Any Swelling; Dose 2 | 37 | 25
  Grade 3 Swelling; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 Swelling; Dose 2 | 1 | 0

5. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited General Symptoms
Description: Assessed solicited general symptoms were meningism and parotid gland swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 meningism and parotid gland swelling = meningism/ parotid gland swelling which prevented normal everyday activities.
Time Frame: Within 43 days (Days 0-42) after each vaccination
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects,with the symptom sheet filled-in.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 330 | 166
Participants
  Any Meningism; Dose 1 | 2 | 1
  Grade 3 Meningism; Dose 1 | 0 | 0
  Any Parotid gland; Dose 1 | 0 | 0
  Grade 3 Parotid gland; Dose 1 | 0 | 0
  Any Meningism; Dose 2: number analyzed (Participants) | 327 | 164
  Any Meningism; Dose 2 | 2 | 0
  Grade 3 Meningism; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 Meningism; Dose 2 | 1 | 0
  Any Parotid gland; Dose 2: number analyzed (Participants) | 327 | 164
  Any Parotid gland; Dose 2 | 0 | 0
  Grade 3 Parotid gland; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 Parotid gland; Dose 2 | 0 | 0

6. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Fever
Description: Any fever was defined as fever greater than or equal to (≥) 38.0 Celsius degrees (°C) and grade 3 fever greater than (>) 39.5°C after vaccination. Related fever was defined as fever assessed by the investigator as related to the vaccination.
Time Frame: Within 43 days (Days 0-42) after each vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 330 | 166
Participants
  Any temperature; Dose 1 | 231 | 104
  Grade 3 temperature; Dose 1 | 54 | 23
  Related temperature; Dose 1 | 160 | 70
  Any temperature; Dose 2: number analyzed (Participants) | 327 | 164
  Any temperature; Dose 2 | 115 | 62
  Grade 3 temperature; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 temperature; Dose 2 | 31 | 13
  Related temperature; Dose 2: number analyzed (Participants) | 327 | 164
  Related temperature; Dose 2 | 29 | 28

7. Secondary Outcome: Number of Subjects Reporting Any (Local or General), Grade 3 and Related Rashes
Description: Rash was defined as: 1) measles/ rubella rashes (macular or maculo-papular rashes): presence of macules, discolored small patches or spots of the skin, neither elevated nor depressed below the skin's surface; 2) varicella rash (maculo-papulo-vesicular): simultaneous presence of macules, papules and vesicles raised above the skin's surface; 3) other types of rash (heat rash, diaper rash etc.). Any rash = occurrence of rash regardless of intensity grade or relationship to vaccination Grade 3 rash ≥ 150 lesions and Related = rash assessed by the investigator as related to the vaccination.
Time Frame: Within 43 days (Days 0-42) after each vaccination
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 330 | 166
Participants
  Any, rash type; Dose 1 | 88 | 42
  Grade 3 rash type; Dose 1 | 9 | 6
  Related rash type; Dose 1 | 37 | 23
  Any, rash type; Dose 2: number analyzed (Participants) | 327 | 164
  Any, rash type; Dose 2 | 40 | 17
  Grade 3 rash type; Dose 2: number analyzed (Participants) | 327 | 164
  Grade 3 rash type; Dose 2 | 6 | 1
  Related rash type; Dose 2: number analyzed (Participants) | 327 | 164
  Related rash type; Dose 2 | 12 | 7

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Event (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any was defined as an adverse event (AE) reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event. Grade 3 was defined as an event that prevented normal activity and Related was defined as an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 43 days (Days 0-42) after first vaccination dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 332 | 166
Participants
  Any AE(s) | 165 | 73
  Grade 3 AE(s) | 8 | 5
  Related AE(s) | 21 | 8

9. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Event (AEs)
Description: as for outcome 8
Time Frame: Within 43 days (Days 86-128) after second vaccination dose
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 332 | 166
Participants
  Any AE(s) | 146 | 76
  Grade 3 AE(s) | 6 | 6
  Related AE(s) | 10 | 6

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed included medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/ incapacity or is a congenital anomaly/ birth defect in the offspring of a study subject.
Time Frame: From first study dose (Day 0) until study end (Week 18)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
Number analyzed (Participants) | 332 | 166
Participants | 27 | 12

ADVERSE EVENTS:
Time Frame: Solicited local symptoms were collected within 4 days after each vaccination.Solicited general symptoms & unsolicited AEs were collected within 43 days after each vaccination. SAEs were collected throughout the entire study period.
Description: The solicited local and general symptoms were only collected for those subjects who filled-in their symptom sheets.
Arm/Group | Priorix-Tetra New WS Group | Priorix-Tetra Current WS Group
All-Cause Mortality (participants affected / at risk) | 0/332 | 0/166
Serious Adverse Events (participants affected / at risk) | 27/332 | 12/166
Other Adverse Events (participants affected / at risk) | 246/332 | 117/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Priorix-Tetra New WS Group (N=332) | Priorix-Tetra Current WS Group (N=166)
Kawasaki's disease (Vascular disorders) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Band neutrophil count increased (Investigations) | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 4 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Testicular retraction (Reproductive system and breast disorders) | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 4 | 4
Acute tonsillitis (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 2 | 2
Bronchopneumonia (Infections and infestations) | 2 | 1
Croup infectious (Infections and infestations) | 2 | 1
Herpangina (Infections and infestations) | 2 | 1
Otitis media acute (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 3 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 1 | 1
Adenovirus infection (Infections and infestations) | 1 | 0
Cellulitis orbital (Infections and infestations) | 0 | 1
Encephalitis viral (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Exanthema subitum (Infections and infestations) | 1 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral rash (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Priorix-Tetra New WS Group (N=332) | Priorix-Tetra Current WS Group (N=166)
Rhinorrhoea; Dose 1 (Respiratory, thoracic and mediastinal disorders) | 31 | 10
Cough; Dose 1 (Respiratory, thoracic and mediastinal disorders) | 24 | 10
Cough; Dose 2 (Respiratory, thoracic and mediastinal disorders) | 24 | 12
Rhinorrhoea; Dose 2 (Respiratory, thoracic and mediastinal disorders) | 24 | 10
Pain; Dose 1 (General disorders) | 62/330 | 28
Redness; Dose 1 (General disorders) | 92/330 | 44
Swelling; Dose 1 (General disorders) | 22/330 | 11
Pain; Dose 2 (General disorders) | 46/327 | 24/164
Redness; Dose 2 (General disorders) | 79/327 | 43/164
Swelling; Dose 2 (General disorders) | 37/327 | 25/164
Diarrhoea; Dose 1 (Gastrointestinal disorders) | 17 | 11
Rash; Dose 1 (Skin and subcutaneous tissue disorders) | 88/330 | 42
Rash; Dose 2 (Skin and subcutaneous tissue disorders) | 40/327 | 17/164
Fever; Dose 1 (Infections and infestations) | 231/330 | 104
Fever; Dose 2 (Infections and infestations) | 115/327 | 62/164
Upper respiratory tract infection; Dose 1 (Infections and infestations) | 50 | 22
Upper respiratory tract infection; Dose 2 (Infections and infestations) | 30 | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.